CLINICAL TRIAL: NCT01084889
Title: National, Multicentre Post-marketing Surveillance Study on Anterior Pelvic Prolapse Reconstruction With Titanium-coated Polypropylene Mesh (TiLOOP® Total 6)
Brief Title: Anterior Pelvic Prolapse Reconstruction With TiLOOP® Total 6
Status: Completed | Type: Observational
Sponsor: pfm medical gmbh (Industry)
Collaborators: Aix Scientifics (Industry); GfE Medizintechnik GmbH (Other); pfm medical titanium gmbh (Unknown); Bayes GmbH (Other); Crolll Gmbh (Other)
Responsible Party: Sponsor
Other Study IDs: pfm 10k001 TiLOOP® Total 6
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Cystocele; Uterine Prolapse
Keywords: polypropylene mesh; Prolapse; Cystocele; Surgical Mesh
MeSH Terms: conditions — Cystocele; Uterine Prolapse; Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- symptomatic genital descensus: Women with a symptomatic genital descensus : at least stage II (ICS-classification according pelvic organ prolapse quanification (POP-Q) system), or stage I with a symptomatic requiring intervention.
  Standard method to implant the TiLOOP® Total 6 surgical mesh transvaginally.
  Interventions: Device: surgical mesh implantation (TiLOOP® Total 6)

INTERVENTIONS:
Device: surgical mesh implantation (TiLOOP® Total 6) — The standard procedure for the surgical repair of anterior prolapse is via the obturator membrane. The surgical mesh TiLOOP® Total 6 is placed transvaginal by the aid of TiLOOP® surgical instruments to place the mesh arms.
  Other Names: TiLOOP® Total 6

SUMMARY:
The purpose of this study is to determine the influence of Anterior Pelvic Prolapse Reconstruction with a titanised polypropylene mesh on rate of erosion and patients quality of live.

DETAILED DESCRIPTION:
This multicentre, non-randomised, observational clinical device investigation will be performed to obtain post-marketing information on the TiLOOP® pelvic floor reconstruction meshes and in particular on the rate of rare erosions of the device under investigation as well as on the improvement of patients' quality of life. It is expected that the rate of erosions is equal or lower compared to competitor devices currently on the market. To verify this, it will be shown that within the first year the erosion rate found for the product under investigation is in the range of 7.9 ± 5.4 %, which is the mean erosion rate found in the recent literature. Erosion, in the sense of the hypothesis, is any erosion 1 requiring more than simply the cut off of a single short filament.

It is also expected that the patient's quality of life is meliorated after implantation of a TiLOOP® Total 6 mesh. To verify this, it will be shown that by means of a validated questionnaire the subjective quality of life after 6 months is significantly better than before implantation.

ELIGIBILITY:
Inclusion Criteria:

* Women with a symptomatic genital descensus : at least stage II (ICS-classification according POP-Q system), or stage I with a symptomatic requiring intervention. This applies to primary as well as recurrent intervention
* Existence of a cystocele.
* Patient is mentally able to understand the nature, aims, or possible consequences of the clinical investigation
* Patient information has been handed out and all written consents are at hand.
* Patient has attained full age.

Exclusion Criteria:

* Pregnancy or unfinished family planning.
* Known intolerance to the mesh-implants under investigation.
* Patients with acute (last 12 months) carcinoma.
* Patients with history of radiotherapy in the pelvic area.
* Genital descensus without any complaints.
* Patients with implanted pelvic floor mesh.
* Systemic steroid treatment.
* Lack of written patients' informed consent.
* Lack of patient compliance regarding data collection, treatment or follow-up investigations in the scope of the protocol.
* Patient is institutionalised by court or official order (MPG §20.3).
* Participation in another clinical investigation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a symptomatic genital descensus treated in the center
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Erosion rate | 12 months
  Erosion, in the sense of the end point, is any erosion requiring more than simply the cut off of a single short filament.
Patient's quality of life | 6 months
  It will be shown that by means of a validated questionnaire whether the subjective quality of life after 6 months is significantly better than before implantation.

SECONDARY OUTCOMES:
Adverse Events | at 6, 12, 36 months
  Documentation and independent evaluation of all complications.
Feasibility of the mesh implantation | 6 months
  Evaluation of questions on usability.
Erosion rate | 36 months
  Erosion, in the sense of the end point, is any erosion requiring more than simply the cut off of a single short filament.
Patient's quality of life | 12 and 36 months
  It will be shown that by means of a validated questionnaire whether the subjective quality of life after 6 months is significantly better than before implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fünfgeld, Dr. MD, Principal Investigator — Klinik Tettnang GmbH, Tettnang
Locations (9):
- Germany (9):
  - Berliner Kontinenzzentrum am Franziskus Krankenhaus,, Berlin
  - Krankenhaus Dresden- Friedrichsstadt, Dresden
  - Evangelisches Diakoniekrankenhaus Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Eppendorf, Hamburg
  - St. Elisabeth Krankenhaus Leipzig,, Leipzig
  - Regionale Kliniken Holding RKH GmbH, Klinikum Ludwigsburg, Ludwigsburg
  - Beckenbodenzentrum München, München
  - Klinik Tettnang GmbH, Tettnang
  - Klinikum Oberlausitzer Bergland gGmbH,, Zittau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Farthmann J, Mengel M, Henne B, Grebe M, Watermann D, Kaufhold J, Stehle M, Fuenfgeld C. Improvement of pelvic floor-related quality of life and sexual function after vaginal mesh implantation for cystocele: primary endpoint of a prospective multicentre trial. Arch Gynecol Obstet. 2016 Jul;294(1):115-21. doi: 10.1007/s00404-016-4014-0. Epub 2016 Jan 18. PMID 26781262
- [Result] Funfgeld C, Stehle M, Henne B, Kaufhold J, Watermann D, Grebe M, Mengel M. Quality of Life, Sexuality, Anatomical Results and Side-effects of Implantation of an Alloplastic Mesh for Cystocele Correction at Follow-up after 36 Months. Geburtshilfe Frauenheilkd. 2017 Sep;77(9):993-1001. doi: 10.1055/s-0043-116857. Epub 2017 Sep 25. PMID 28959063
- See also: Quality of life and pelvic organ prolapse-related symptoms after pelvic floor reconstruction with a titanized polypropylene mesh for cystocele: long-term results in a 36 month follow-up by Fünfgeld et al, 2018 — http://www.pelviperineology.org/december-2018/pdf/pelviperineology-december-2018.pdf